CLINICAL TRIAL: NCT00114010
Title: Phase 1 Study of the Safety of Immunization of Naive Individuals With AMA1-C1/Alhydrogel [R], an Asexual Blood-Stage Vaccine for Plasmodium Falciparum Malaria, and the Effect of Immunization on Antigen-specific Memory and Plasma B Cells and T Cells
Brief Title: Experimental Vaccine for Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 050133; 05-I-0133
Record Dates: First submitted 2005-06-11; First posted 2005-06-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-08-19

CONDITIONS: Malaria
Keywords: B Cells; T Cells; Erythrocyte Stage; Antibody; Immunogenicity; Healthy Volunteer
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Drug: AMA1/Alhydrogel

SUMMARY:
This study will examine the safety and immune response of healthy adult volunteers to AMA1-C1, an experimental malaria vaccine developed by the NIAID. Malaria affects about 300 million to 500 million people worldwide each year, causing from 2 million to 3 million deaths. Increasing drug resistance to the malaria parasite, as well as widespread resistance of mosquitoes (the insects that transmit the parasite) to pesticides are reducing the ability to control malaria through these strategies. A vaccine that could reduce illness and death from malaria would be a valuable new resource in the fight against this disease. Early tests of AMA1-C1 in 66 people in the United States and in Mali, West Africa, found no serious side effects of the vaccine. This study will test a shorter schedule of vaccinations with AMA1-C1 than that used in the previous studies.

Healthy volunteers between 18 and 50 years of age who weigh at least 110 pounds and with no travel to malaria endemic areas in the past 12 months may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, and a urine pregnancy test for women who are able to bear children.

Participants are randomly assigned to receive three injections of either the experimental malaria vaccine or a placebo (a solution that does not contain the vaccine) over a 2-month period. The shots are given in an upper arm muscle, each 1 month apart. On the day of each injection, participants give a history of symptoms since the last visit, have a brief physical examination and blood test and, for women, a blood or urine pregnancy test. After the injection, participants remain in the clinic 60 minutes for observation. In addition to the injections, participants undergo the following procedures:

* Record temperature and symptoms on a diary card daily for the first 7 days after each injection.
* Follow-up clinic visits 1, 3, 7 and 14 days after each shot to check for side effects. Blood samples are drawn before each injection and at each return clinic visit to check the safety and immune response to the vaccine.
* Have apheresis, a special procedure that separates certain components of the blood, 7 days after each injection to measure the function of germ-fighting blood cells. For this procedure, blood is drawn through a needle in an arm vein and directed into a machine that separates the different types of blood cells. The white cells are collected in a plastic ...

DETAILED DESCRIPTION:
The study is a randomized, single-blinded (blinded to volunteers) placebo-controlled Phase 1 clinical trial in healthy adult volunteers designed to evaluate the safety and reactogenicity of a new malaria blood stage vaccine candidate, and to elucidate the immunogenicity of the antigen, AMA1-C1, formulated on Alhydrogel [R]. The trial will last 42 weeks. Volunteers will be recruited and screened, and those determined to be eligible will be enrolled in the study, based on the inclusion and exclusion criteria described in Section 4.0 in this protocol. After providing written informed consent the volunteers will be enrolled and randomly allocated to receive 80 microgram dose of AMA1-C1 formulated on Alhydrogel [R] (12 volunteers) or Alhydrogel [R] alone (6 volunteers) at 0, 1 and 2 months. After each injection, volunteers will be observed for 60 minutes for immediate reactions. Volunteers will return to the clinic on study days 1, 3, 7, and 14 following each injection for clinical assessment and collection of blood samples for evaluation of immune responses. Leukaphereses will be performed 7 days after the third vaccination to obtain peripheral blood mononuclear cells for B and T cell studies. Safety data for the cohort up to and including follow up day 14 after the first, second and third injection will be available for review by the Medical Monitor.

Immunogenicity of the vaccine will be assessed by standardized assays for antibody levels against AMA1-3D7 and AMA1-FVO, and an in vitro growth inhibition assay (GIA). The cellular basis of the immune responses will be evaluated by enumeration of relevant B and T cell subpopulations, including total and antigen-specific naive, memory and effector subpopulations specific for the antigens. The frequencies of B and T cells specific for the vaccine antigens in the group that received AMA1-C1/ Alhydrogel [R] will be compared to those in the group receiving Alhydrogel [R] alone. The total and antigen-specific cell frequencies in pre-immune (day 0) samples will serve as additional negative controls for the immunization. The goal of the study is to augment previously collected safety data for the 80 microgram antigen dose with a larger cohort, and to study the safety and immunogenicity of an accelerated vaccination schedule.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males or females between 18 and 50 years, inclusive.

Available for the duration of the trial (34 weeks)

Willingness to participate in the study as evidenced by signing the informed consent document.

Weighing at least 110 pounds.

EXCLUSION CRITERIA:

Age less than 18 years because insufficient data are available in adults to judge potential risk in children.

Pregnancy as determined by a positive urine Beta-hCG (if female).

Participant unwilling to use reliable contraception methods (condoms or oral contraceptives) for the duration of the trial (if female).

Currently lactating and breast-feeding (if female).

Participant unwilling to undergo apheresis.

Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.

Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.

Laboratory evidence of liver disease (aspartate aminotransferase AST greater than the upper limit of normal of the testing laboratory and/or total bilirubin levels greater than the upper limits of normal of the testing laboratory).

Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory).

Laboratory evidence of hematologic disease (absolute neutrophil count less than 1,500/mm(3); hemoglobin less than the lower limit of normal of the testing laboratory, by sex; or platelet count less than 140,000/mm(3).

Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Participation in another investigational vaccine or drug trial within 30 days of enrolling in this study, or while this study is ongoing.

Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.

History of a severe allergic reaction or anaphylaxis to drugs or foods.

Asthma that has resulted in an emergency room visit or hospitalization within the last 6 months.

Positive ELISA and confirmatory Western blot tests for HIV-1.

Positive ELISA and standard confirmatory tests for HCV.

Positive HBsAg by ELISA.

Known immunodeficiency syndrome.

Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of enrolling in this study or while the study is ongoing.

Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.

History of a surgical splenectomy.

Receipt of blood products within the past 6 months.

Previous receipt of an investigational malaria vaccine.

Receipt of antimalarial prophylaxis during the past 12 months.

Prior malaria infection.

Travel to a malaria-endemic country during the past 12 months or planned travel to a malaria-endemic country during the course of the study.

History of a known allergy to nickel.

History of known allergy to yeast.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2005-04-01; Primary Completion 2006-12-22 (Actual); Study Completion 2006-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Good MF, Kaslow DC, Miller LH. Pathways and strategies for developing a malaria blood-stage vaccine. Annu Rev Immunol. 1998;16:57-87. doi: 10.1146/annurev.immunol.16.1.57. PMID 9597124
- [Background] Narum DL, Thomas AW. Differential localization of full-length and processed forms of PF83/AMA-1 an apical membrane antigen of Plasmodium falciparum merozoites. Mol Biochem Parasitol. 1994 Sep;67(1):59-68. doi: 10.1016/0166-6851(94)90096-5. PMID 7838184
- [Background] Crewther PE, Culvenor JG, Silva A, Cooper JA, Anders RF. Plasmodium falciparum: two antigens of similar size are located in different compartments of the rhoptry. Exp Parasitol. 1990 Feb;70(2):193-206. doi: 10.1016/0014-4894(90)90100-q. PMID 2404781